CLINICAL TRIAL: NCT04762251
Title: What Or When to Eat to Reduce the Risk of Type 2 Diabetes (WOW)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Adelaide (Other)
Collaborators: Australian Catholic University (Other); La Trobe University (Other)
Responsible Party: Principal Investigator, A/Prof Leonie Heilbronn, Group Leader, Obesity and Metabolism, University of Adelaide
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 14023
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Time-restricted Eating; Diet Quality
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time-restricted eating (TRE) (Experimental): The TRE group will be instructed to follow TRE (9 h/day) every day for 12 months with no other dietary instructions or advice provided. The TRE group will attend the same consult schedule as the CP group, but consultations will focus on timing of dietary intake and strategies to promote adherence. No dietary guidance regarding quantity or quality will be provided. Participants will be able to self-select the precise 9-h schedule that will best suit their lifestyles, with the caveat that the latest time of eating will be set at 7:00 pm. Outside of the elected eating window, participants will be allowed to consume water and black coffee and/or tea.
  Interventions: Other: Time-restricted eating
- Current Best Practice (CP) (Active Comparator): This group is designed to act as a comparator using 'standard care' in dietetics practice. Dietary advice provided to this participant group will be performed by Accredited Practicing Dietitians (APDs) in line with evidence-based guidelines, specifically the T2DM best-practice guidelines plus Australian Dietary Guidelines (i.e. Australian Guide to Healthy Eating) to improve diet quality, and strategies to promote adherence. No specific advice will be provided regarding time of day to start and finish eating and/or drinking (since this information is not outlined in current practice guidelines).
  Interventions: Other: Current Best Practice

INTERVENTIONS:
Other: Time-restricted eating — Time restricted eating for a self-selected 9 hour window per day
  Arms: Time-restricted eating (TRE)
Other: Current Best Practice — Best practice guidelines to improve diet quality
  Arms: Current Best Practice (CP)

SUMMARY:
A parallel, single-blinded, multi-centre randomized controlled trial conducted at the South Australian Health and Medical Research Institute (SAHMRI) and the Mary Mackillop Institute for Health Research (MMIHR; Australian Catholic University), by researchers from the University of Adelaide, Australian Catholic University and La Trobe University.

DETAILED DESCRIPTION:
In a parallel groups design, a total of 268 individuals will be recruited across both sites. After a 2-week baseline period, and a baseline metabolic visit, participants will be randomized into one of two groups (TRE, time-restricted eating; CP, current practice guidelines). All participants will receive five (5) telehealth consultations at baseline, week 2, 4, 8 and 12, the content of which will be based around their randomized condition. They will undergo metabolic testing on two (2) further occasions (4 months, 12 months) over a 12-month period to assess the changes in primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Study participants will be aged 35 to 70 years, overweight or obese (BMI: >25 but <45 kg/m2), ≥15 on the AUSDRISK assessment tool and have HbA1c <6.5% at screening

Exclusion Criteria:

Type 1 or type 2 diabetes, or diabetes detected at screening HbA1c ≥6.5% (48 mmol/mol).

* A personal history/diagnosis (self-reported) of:

  * major psychiatric disorders (schizophrenia, major depressive disorder, bipolar disorder, eating disorders)
  * gastrointestinal disorders/disease (including malabsorption)
  * haematological disorders (i.e. thalassemia, iron-deficiency anaemia)
  * insomnia
  * currently receiving, or have received treatment/diagnosis of cancer in the past 3 years (excluding non-melanoma skin cancer)
  * significant liver or kidney disease
  * previous or planned gastro-intestinal surgery (including bariatric surgery)
  * Congestive heart failure (NYHA stage 2 or above)
  * Previous myocardial infarction or significant cardiac event ≤ 6 months prior to screening
  * Previous cerebrovascular event ≤ 12 months prior to screening

and/or any other condition deemed unstable by the study physician.

Currently taking the following medications:

* any medication used, or known to lower blood glucose, or antidiabetic medications, including, but not limited to: SGLT2 inhibitors, metformin, sulfonylureas, glucagon-like peptide-1 (GLP-1) analogues [i.e. exenatide], thiazolidinediones or DPP-IV inhibitors [i.e. 'gliptins'])
* Medications affecting weight, appetite or gut motility, including, but not limited to: (domperidone, cisapride, orlistat, phentermine, topiramate).
* Diuretics (i.e. frusemide, thiazides) or combination blood pressure medications containing a diuretic
* Beta-blockers
* Glucocorticoids
* Anti-epileptic medications
* Antipsychotic medications
* Opioid medications unless combined with paracetamol in a single formulation and used occasionally on a PRN basis

Additional exclusion criteria include:

* do not consume a regular breakfast (i.e. eat breakfast on an average of 5 or more days per week), and do not eat for more than 12 hours per day on an average of 5 or more days per week
* have an extreme or restricted pattern of eating (i.e. following an intermittent fasting diet) or are already engaged in a TRE protocol
* shift-workers
* pregnant, planning a pregnancy or currently breastfeeding
* those who have lost or gained >5% of body weight in the last 6 months
* current smokers of cigarettes/marijuana/e-cigarettes/vaporisers
* anyone unable to comprehend the study protocol or provide informed consent (i.e. due to English language or cognitive difficulties)
* Participants will not have seen a dietitian in the preceding 3 months.
* score on K10 ≥30 (Kessler Psychological Distress scale)
* score on EDEQ ≥2.8 (Eating Disorder Examination Questionnaire)

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
HbA1c | baseline, 4 months
  Glycated haemoglobin concentration

SECONDARY OUTCOMES:
HbA1c | 12 months
  Glycated haemoglobin concentration
Fasting blood glucose | baseline, 4 months, 12 months
  fasting blood glucose concentrations
Fasting insulin | baseline, 4 months, 12 months
  fasting insulin concentrations
HOMA-IR | baseline, 4 months, 12 months
  HOMA-IR
Nocturnal glucose | baseline, 4 months
  AUC of glucose assessed by CGM from midnight to 0400

OTHER OUTCOMES:
Per protocol analysis | 4 months, 12 months
  Per protocol analysis of data from participants who self-report adherence as 5-6 days per week or every day at 3.5 and 4 month adherence questionnaires ("adherent to the protocol")
Body weight | baseline, 4 months, 12 months
  body weight (assessed after an overnight fast, in a hospital gown)
Body composition | baseline, 4 months, 12 months
  components of body composition assessed by DXA: fat mass (as percent body fat and kg), fat free mass (FFM, kg), visceral adipose tissue (VAT, g) and bone mass (kg)
Waist circumference | baseline, 4 months, 12 months
  waist circumference (cm)
Hip circumference | baseline, 4 months, 12 months
  hip circumference (cm)
Blood lipids | baseline, 4 months, 12 months
  total, HDL and LDL cholesterol and triglycerides
hs-CRP | baseline, 4 months, 12 months
  high sensitivity C-reactive protein (hs-CRP)
Liver markers | baseline, 4 months, 12 months
  alanine transaminase (ALT) and aspartate aminotransferase (AST)
24h assessment of glycaemia | baseline, 4 months
  24h glucose measures assessed by CGM (including, but not limited to, time in range, CV)
Physical activity | baseline, 4 months, 12 months
  Components of activity (Step count, time in bed) assessed by inclinometer
Sleep duration | baseline, 4 months, 12 months
  Sleep duration calculated from self-reported sleep/wake times
Cardiovascular measures | baseline, 4 months, 12 months
  blood pressure and heart rate assessed using automated sphygmomanometer
meal timing / eating window | baseline, 4 months, 12 months
  duration of eating window and individual meal times calculated from time-stamped food photos and/or self-reported meal times
Dietary intake | baseline, 4 months, 12 months
  energy and macronutrient composition calculated from food diaries (research food diary app)
Adherence | 3.5, 4, 11.5, 12 months
  measures of adherence assessed by self-report (questionnaire)
Chronotype | baseline, 3.5, 4, 11.5, 12 months
  participant chronotype calculated from MEQ-SA questionnaire
TRE vs CP on ambulatory blood pressure and renal function (sub-study) | baseline, 4 months
  Day and night time blood pressure (systolic, diastolic), dipping, morning surge, heart rate, blood pressure and heart rate variability. mesor, phase and amplitude of 24 hour ambulatory blood pressure monitoring; change in eGFR, creatinine, albumin urinary albumin:creatinine ratio, blood urea nitrogen and C-RP
TRE vs CP on CGM outcomes in a subset of individuals with pre-diabetes (sub-study) | 4 months, 12 months
  Change in CGM metrics (including 2 hour at-home glucose challenge) in participants with HbA1c >5.7% at baseline
TRE vs CP on quality of life, mood, sleep and food preferences (sub-study) | 4 months, 12 months
  Assessment of lifestyle using AQOL, mood using DASS-21 and CIA, sleep using PSQI and food preferences using NQOL and DRQOL
TRE vs CP on diet quality (sub-study) | 4 months, 12 months
  Assessment of changes in diet quality in TRE vs CP groups over 12 months using HEIFA (Healthy eating index for Australian Adults)
TRE vs CP on barriers and enablers of adherence (sub-study) | 4 months, 12 months
  Qualitative interview of a subset of participants to identify barriers and enablers of adherence to TRE vs CP advice

CONTACTS AND LOCATIONS:
Overall Officials: Leonie Heilbronn, PhD, Principal Investigator — University of Adelaide; John Hawley, PhD, Principal Investigator — Australian Catholic University
Locations (2):
- Australia (2):
  - South Australian Health and Medical Research Institute, Adelaide, South Australia
  - Mary Mackillop Institute for Health Research, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study will be available from the corresponding author for a period of 36 months from publication, upon reasonable request for academic use. The data will not be made publically available, as it contains information that could compromise research participant consent.
Supporting Information: Study Protocol, SAP
Time Frame: 36 months from date of publication
Access Criteria: Reasonable requests of data for academic use will be considered. Requests can be made to the corresponding author of the publication. Data will not be made publically available as it contains information that could compromise research participant consent.

REFERENCES:
- [Derived] Charrouf R, Parr EB, Hutchison AT, Flint SA, Teong XT, Wittert G, Vincent AD, Brennan L, Devlin BL, Hawley JA, Heilbronn LK. Effect of time restricted eating versus current practice in dietetics on glycaemic control and cardio-metabolic outcomes in individuals at risk of developing type 2 diabetes: Protocol for a multi-centre, parallel group, non-inferiority, randomised controlled trial. Contemp Clin Trials. 2024 Nov;146:107696. doi: 10.1016/j.cct.2024.107696. Epub 2024 Sep 17. PMID 39299545
- See also: preprint of the study protocol — https://papers.ssrn.com/sol3/papers.cfm?abstract_id=4788134

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-02-29): https://cdn.clinicaltrials.gov/large-docs/51/NCT04762251/SAP_000.pdf